CLINICAL TRIAL: NCT07287475
Title: Application of Growth Factors Derived From Platelets to Accelerate Healing and Reduce Post-extraction Complications in Diabetic Individuals
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Amal Jamjoom, BDS, MS., Assistant Professor at KAU, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 264-12-23
Record Dates: First submitted 2025-12-01; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Diabete Mellitus
Keywords: Diabetic; A-PRF; Extraction; Socket
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPRF (Other): Experimental: A- PRF in Extraction sockets in Diabetic patients. Arm Description: A randomized, double-blinded, split-mouth clinical trial was conducted at King Abdulaziz University Dental Hospital. Diabetic patients requiring bilateral extraction of the same tooth were enrolled. One socket was randomly assigned to receive A-PRF while the contralateral socket served as the control. Healing was assessed using digital intraoral scanning at baseline, 1 week, and 2 weeks post-extraction.
  Interventions: Procedure: Platelet rich fibrin
- Control (No Intervention): Nothing was placed in the socket

INTERVENTIONS:
Procedure: Platelet rich fibrin — Description: A-PRF is a biologically active scaffold that fits into the proven principles of the physiology of the wound-healing process. Its action lies in the controlled and prolonged release of fundamental factors like the PDGF (platelet-derived growth factor), TGF-β (transforming growth factor beta), and VEGF (vascular endothelial growth factor) which collectively enhance cellular migration, angiogenic events, and extracellular matrix remodeling factors of repair in the recovery of the tissues.
  Arms: iPRF

SUMMARY:
To evaluate soft tissue closure in diabetic extraction sockets using digital scans.

To compare healing between sockets treated with Advanced Platelet Rich Fibrin (A-PRF) vs. untreated control sites.

To assess post-operative discomfort and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years or older
* Need bilateral tooth extraction
* Sockets should be the same size
* Diabetic/ uncontrolled
* No other disease
* Non- smoker
* Non-pregnant or lactating female

Exclusion Criteria:

* Patients below 18 years
* Patients with diseases different from diabetes
* Bleeding disorders
* Pregnancy
* Lactation,
* Tobacco use (conventional or electronic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Socket size | 3 weeks
  Soft tissue healing of extraction sockets

CONTACTS AND LOCATIONS:
Locations (1):
- King AbdulAziz University, Jeddah, Mekkah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] 1. Alwin Robert, A. and M.A. Al Dawish, Microvascular complications among patients with diabetes: An emerging health problem in Saudi Arabia. Diab Vasc Dis Res, 2019. 16(3): p. 227-235. 2. Kudiyirickal, M.G. and J.M. Pappachan, Diabetes mellitus and oral health. Endocrine, 2015. 49(1): p. 27-34. 3. Mohseni Homagarani, Y., et al., The effect of diabetes mellitus on oral health-related quality of life: A systematic review and meta-analysis study. Front Public Health, 2023. 11: p. 1112008. 4. Davis, V.L., et al., Platelet-rich preparations to improve healing. Part I: workable options for every size practice. J Oral Implantol, 2014. 40(4): p. 500-10. 5. Singh, N., D.G. Armstrong, and B.A. Lipsky, Preventing foot ulcers in patients with diabetes. Jama, 2005. 293(2): p. 217-28. 6. Al-Rubeaan, K., et al., Diabetic foot complications and their risk factors from a large retrospective cohort study. PLoS One, 2015. 10(5): p. e0124446. 7. Yoo, J.J., et al., The effect of diabetes on tooth loss caused by periodontal disease: A nationwide population-based cohort study in South Korea. J Periodontol, 2019. 90(6): p. 576-583. 8. Wang, Q., et al., Clinical analysis of medication related osteonecrosis of the jaws: A growing severe complication in China. J Dent Sci, 2018. 13(3): p. 190-197. 9. Ribeiro, L.M., et al., Streptococcus anginosus and Phalangeal Osteomyelitis: An Unusual Presentation. J Orthop Case Rep, 2020. 10(9): p. 19-22. 10. Gholinejad Ghadi, N., et al., [Not Available]. J Mycol Med, 2018. 28(2): p. 399-402. 11. Zhou, S., et al., The role of IFT140 in early bone healing of tooth extraction sockets. Oral Dis, 2022. 28(4): p. 1188-1197. 12. de Sousa Gomes, P., et al., Molecular and Cellular Aspects of Socket Healing in the Absence and Presence of Graft Materials and Autologous Platelet Concentrates: a Focused Review. J Oral Maxillofac Res, 2019. 10(3): p. e2. 13. Takahashi, S., et al., Lymphangiogenesis and NOS Localization in Healing Process

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT07287475/Prot_SAP_000.pdf